CLINICAL TRIAL: NCT05933018
Title: Interconnection Between Night Hyperglycemia and Fatty Liver in Type 1 Diabetes Mellitus
Brief Title: Night Hyperglycemia and Fatty Liver in Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Elena Chertok, MD, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0101-22-EMC
Record Dates: First submitted 2023-06-18; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Type1diabetes; Fatty Liver
Keywords: Type 1 diabetes
MeSH Terms: conditions — Fatty Liver; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- type 1 diabetes (Other): patients with type 1 diabetes underwent liver elastography
  Interventions: Diagnostic Test: liver elastography

INTERVENTIONS:
Diagnostic Test: liver elastography — the imaging of the liver will perform in the fasting state, in the morning hours by one specialist, dedicated to this procedure,

SUMMARY:
This clinical trial aims to discover the relationship between hyperglycemia at night and early morning hours and the presence of fatty liver in patients with type 1 diabetes.

The main question it aims to answer are:

• if hyperglycemic patterns related to metabolic parameters in type 1 diabetes The data from the insulin pump and sensor will be processed. The patients will be divided into two groups. One group without night hyperglycemia and the other with night hyperglycemia. Investigators will perform liver elastography for these two groups. The presence or absence of hepatic steatosis will be evaluated in these groups according to the data.

DETAILED DESCRIPTION:
Introduction Normal subjects have well-defined 24-hour cycles of insulin secretion and plasma insulin levels (rising in the early morning, peaking in the afternoon, and declining at night.

The dawn phenomenon is the result of an exaggeration of the physiologic impairment of insulin sensitivity was noted during the early morning hours. During previous studies, no exact explanation of this phenomenon was found. According to the studies, high growth hormone levels with decreased suppression by hyperglycemia, central hypersensitivity to growth hormone-releasing hormone (GHRH), low insulin-like growth factor-I (IGF-I), high insulin-like growth factor-binding protein-1 (IGFBP-1), and peripheral resistance to growth hormone are involved in the pathogenesis of Dawn syndrome. The etiology, prevalence, and consequences of hepatic steatosis in type 1 diabetes remain poorly understood.

Methods The study will include 120 consecutive patients with type 1 diabetes, using an insulin pump and continuous glucose monitoring device treated in our clinic. Investigators will extract the data related to glucose levels and pump programming. The data about glucose levels and insulin requirements during the night hours will be collected. The study participants will be divided into two groups according to the presence or absence of night hyperglycemia. We will perform liver elastography on 100 study patients.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes patients
* C- PEPTIDE level <0.6
* continuous glucose monitoring system
* insulin pump users

Exclusion Criteria:

* pregnancy
* type 2 diabetes
* non-pump or sensor users
* unwilling to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
to evaluate presence of fatty liver in type 1 diabetes | through study completion, an average of 1 year.
  Liver fat and fibrosis will be assessed by controlled attenuation parameter (CAP) and liver stiffness measurements (LSM) by FibroScan . The attenuation parameter ( CAP ) >270 db/m will be consistent with fatty liver and liver stiffness > 7 will be consistent with liver fibrosis

SECONDARY OUTCOMES:
presence of metabolic syndrome in type 1 Diabetes Mellitus | through study completion, an average of 1 year
  presence of metabolic syndrome in patients with type 1 diabetes including elevated BMI, increased waist circumference, presence of elevated triglycerides, presence of hypertension will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Elena Chertok Shacham, MD, Principal Investigator — Emek Medical Center
Locations (1):
- Emek Medical Center, Afula, Israel/zaphon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Memaj P, Jornayvaz FR. Non-alcoholic fatty liver disease in type 1 diabetes: Prevalence and pathophysiology. Front Endocrinol (Lausanne). 2022 Dec 1;13:1031633. doi: 10.3389/fendo.2022.1031633. eCollection 2022. PMID 36531463